CLINICAL TRIAL: NCT07317349
Title: The Effect of a Continuous 1-Hour Time Delay on Circadian Rhythms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Independent Research Fund Denmark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1-10-72-143-25; 10.46540/425600108B (Other Grant/Funding Number: Independent Research Fund Denmark)
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Circadian Rhythms; Time Perception; Sleep
Keywords: circadian phase delay; Healthy adults

STUDY DESIGN:
Intervention Model Description: Participating couples will need to live in this environment for 5 consecutive days. By lottery draw, you as a couple will either be exposed to a fixed daily routine, where all activities occur at the same time every day, or a daily time delay of 1 hour, where all activities will be delayed by one hour.
Masking Description: Open-label, single-group basic science study; no masking used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed daily routine (Experimental): All activities occur at the same time every day. During the five days, participants will have to complete various daily tests and also be asked to provide 8 saliva samples during days 1, 3, and 5
  Interventions: Behavioral: Fixed daily routine
- Daily time delay of 1 hour (Experimental): All activities will be delayed by one hour. During the five days, participants will have to complete various daily tests and also be asked to provide 8 saliva samples during days 1, 3, and 5
  Interventions: Behavioral: Daily time delay

INTERVENTIONS:
Behavioral: Fixed daily routine — All activities occur at the same time every day
  Arms: Fixed daily routine
Behavioral: Daily time delay — All activities will be delayed by one hour per day over a 5 day period.
  Arms: Daily time delay of 1 hour

SUMMARY:
The purpose of this study is to investigate whether the experience of a daily time delay can affect our internal circadian rhythm.

ELIGIBILITY:
Inclusion Criteria

* Healthy adults aged 23-45 years
* Part of a heterosexual, cohabiting couple willing to participate together in a five-day in-laboratory study
* Both partners meet all inclusion criteria
* Completion of at least upper-secondary education
* Maintain a regular sleep-wake schedule
* Habitual sleep timing within a normative range (non-extreme chronotype), assessed using the Morningness-Eveningness Questionnaire (MEQ) or the Munich Chronotype Questionnaire (MCTQ)
* Both partners fall within the acceptable chronotype range to ensure aligned sleep-wake patterns
* Low seasonality scores on the Seasonal Pattern Assessment Questionnaire (SPAQ)
* Free from underlying sleep or mood disorders

Exclusion Criteria

* Engages in night-shift work or maintains an irregular work or sleep schedule
* International travel involving a time-zone change of more than two hours within the past two months, or anticipated travel before study completion
* Diagnosed neurological, psychiatric, or sleep disorder (e.g., insomnia, sleep apnea, bipolar disorder)
* High risk of sleep apnea, defined as a Berlin Questionnaire score >2 (Lauritzen et al., 2018)
* Use of medications known to affect sleep, alertness, melatonin secretion, or circadian timing
* Unable or unwilling to comply with behavioral restrictions, including refraining from electronic devices displaying time cues unless clocks are removed and devices are disconnected from Wi-Fi
* Unable or unwilling to comply with consumption restrictions, including abstaining from caffeine, alcohol, and melatonin-rich foods during the study
* Extreme chronotype, defined as a habitual midsleep time outside 03:00-05:00 on the MCTQ or classification as an extreme morning or extreme evening type on the MEQ
* Daily caffeine consumption exceeding 400 mg (approximately 4-5 cups of coffee)
* Current smoker or smoking within the past six months

Ages: 23 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Phase shift in circadian rhythm markers | Comparing samples on days 1, 3, 5
  The primary outcome is the timing of dim light melatonin onset, a marker of circadian phase. Saliva samples will be collected at regular intervals under dim light, and the time when melatonin exceeds 3 pg/mL will be recorded for each participant. This allows measurement of circadian phase shifts across conditions.

SECONDARY OUTCOMES:
Psychomotor Vigilance Task (PVT) Median Reaction Time | Performance will be measured at regular intervals on days 1 - 5 to track changes over the course of the study.
  Median reaction time (milliseconds) on a brief psychomotor vigilance task (PVT) six times each day. Participants respond as quickly as possible to visual stimuli presented at random inter-stimulus intervals. For each block, the median reaction time is computed; additional indices such as lapses (responses > 500 ms) may be derived. Changes in PVT performance across the the 5 days are analysed in relation to circadian phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Department of Psychology and Behavioural Sciences, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the published results will be shared with other researchers upon reasonable request, in accordance with Danish data protection regulations, institutional policies, and ethics approval. Data will be pseudonymised before sharing and no direct identifiers (e.g., name, contact details, personal ID numbers) will be included. Any data elements that could reasonably lead to re-identification in combination with other information will be removed or aggregated where necessary.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: De-identified individual participant data and supporting documents will be made available beginning within 12 months after publication of the main results article and will remain available for at least 5 years thereafter.
Access Criteria: De-identified individual participant data (IPD), together with the study protocol, statistical analysis plan, and analytic code, will be available to qualified researchers affiliated with recognised research institutions who submit a methodologically sound proposal and obtain any required ethical or institutional approvals. Requests should describe the planned analyses and data needed. Approved requesters will sign a data use agreement prohibiting re-identification of participants and requiring appropriate data security. Data will be shared via secure transfer or a controlled-access repository approved by Aarhus University.

REFERENCES:
- See also: Sleep & Circadian Psychology Research Unit - Aarhus University (information on research in sleep, circadian rhythms) — https://psy.au.dk/en/circadianpsychology